CLINICAL TRIAL: NCT05898503
Title: Effects of Different Types of Exercise on Cognitive Function in Postmenopausal Hypertensive Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EODTOEOCFIPHW
Record Dates: First submitted 2023-04-20; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-04

CONDITIONS: Cognitive Function; Hypertension
Keywords: Exercise intervention; Postmenopausal; Cognitive function; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Resistance Training; Health Promotion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Combined training group (Experimental)
  Interventions: Behavioral: Walking exercise + resistance training
- Resistance training group (Experimental)
  Interventions: Behavioral: Resistance training
- Walking exercise group (Experimental)
  Interventions: Behavioral: Walking exercise
- Positive control group (Active Comparator)
  Interventions: Behavioral: Health promotion
- Negative control group (Sham Comparator)
  Interventions: Behavioral: Health promotion

INTERVENTIONS:
Behavioral: Walking exercise + resistance training — Walking exercise and resistance training for 12 weeks
  Arms: Combined training group
Behavioral: Resistance training — Resistance training for 12 weeks
  Arms: Resistance training group
Behavioral: Walking exercise — Walking exercise for 12 weeks
  Arms: Walking exercise group
Behavioral: Health promotion — Health promotion for 12 weeks
  Arms: Negative control group; Positive control group

SUMMARY:
Brief Summary: The study was conducted in two parts, the first of which was carried out using a cross-sectional design approach to explore the relationship between cognitive function and autonomic function, brain function, inflammation and oxidative stress, vascular function, fitness levels, cardiorespiratory endurance and lipid metabolism. The second part uses a repeated measures design approach in a randomised controlled design to explore the effects of different types of exercise on cognitive decline in postmenopausal hypertensive women and their mechanisms of action.

DETAILED DESCRIPTION:
Detailed Description: The study was conducted in 2 parts. Part I: was conducted using a cross-sectional design approach to explore the relationship between cognitive function and autonomic function, brain function, inflammation and oxidative stress, vascular function, fitness levels, cardiorespiratory endurance and lipid metabolism. Multiple linear regression was used to analyse the multiple linear relationships between changes in cognitive function and the above influences. Multiple logistic regression analysis was also used to analyse which of the above risk factors might be independent predictors of cognitive decline. Therefore, a combination of both regression analyses was used to further explore the multiple linear relationships between cognitive function and the aforementioned influencing factors, providing a viable causal and theoretical basis for the next exercise intervention.

The second part of the study is to test the viability of the vascular function theory. The "vascular function theory" refers to the use of exercise to improve aerobic capacity, improve blood circulation to the heart, and improve cerebrovascular function, which in turn improves cognitive function. Based on the above hypothesis, this study aims to investigate the possible effects of 12 weeks of different types of exercise on cognitive decline in post-menopausal women with HTN, and to lay the theoretical and practical foundation for the extension of the exercise intervention to other ages and populations.

ELIGIBILITY:
1. postmenopausal HTN women aged 55 to 65 years
2. 140 mm Hg ≤ SBP < 160 mm Hg) and/or 90 mmHg < DBP < 99 mmHg (2016 edition of the Chinese guidelines for hypertension control)
3. non-persistent hypertension (i.e., continuous use of three or more antihypertensive drugs and blood pressure still within the normal range, or continuous use of four or more antihypertensive drugs to control blood pressure
4. no other metabolic and cardiovascular problems
5. able to participate in physical activity
6. no exercise habit (no more than 6,000 steps per day)
7. alcohol and smoking prohibited
8. moderate risk classification of having cardiovascular disease
9. voluntary participation

Exclusion criteria:

1 pre-menopausal, not falling under the above conditions 2 blood pressure not exceeding the above range 3 refractory hypertension and secondary hypertension 4 metabolic and cardiovascular diseases 5 unable to exercise for their own reasons 6 regular exercise (more than 6,000 steps per day) 7 poor lifestyle habits such as alcohol and smoking 8 suffering from cardiovascular disease risk classification of high or low

b.

Inclusion criteria for the negative control group:

1. postmenopausal women aged 55 to 65 years
2. SBP ≥ 120 mmHg, DBP < 90 mmHg
3. good physical condition
4. practice daily exercise (more than 6000 times daily)
5. do not drink or smoke
6. have a risk classification of no risk for cardiovascular disease
7. voluntary participation

Exclusion criteria:

1. pre-menopausal and not in the above category
2. SBP and DBP values below normal
3. general health, disability or other medical conditions
4. poor diet, alcohol abuse, smoking, etc.
5. no low risk cardiovascular risk classification

Ages: 55 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2023-04-23 (Actual); Primary Completion 2024-04-23 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
MOCA score | 12 weeks
  The change of MOCA score. Montreal cognitive assessment (MoCA). The MoCA scale includes cognitive functions such as visuospatial and executive functions, naming, attention, language, abstraction, delayed recall and orientation, and evaluates the level of cognitive function from several cognitive dimensions. The MoCA has a total score of 30 questions, with 26 being normal and <26 being cognitive decline.

SECONDARY OUTCOMES:
Blood pressure | 12 weeks
  The change of blood pressure before and after intervention.
Quiet heart rate | 12 weeks
  The change of quiet heart rate before and after intervention.
Waist and hip circumference | 12 weeks
  The change of waist circumference and hip circumference before and after intervention.
Body fat percentage | 12 weeks
  The change of body fat percentage before and after intervention.
Lipid metabolism indicators | 12 weeks
  The change of lipid metabolism indicators before and after intervention. Lipid metabolism indicators include: total cholesterol (TC), triglycerides (TG), high-density lipoprotein cholesterol (HDL-C) and low-density lipoprotein cholesterol (LDL-C).
Cardiorespiratory endurance indicator | 12 weeks
  The change of cardiopulmonary endurance indicator before and after intervention. Cardiopulmonary endurance indicator: maximal oxygen uptake (VO2max) was determined using exercise cardiorespiratory testing system.
Serum interleukin-6 (IL-6) | 12 weeks
  The change of inflammation indicators before and after intervention.
High-sensitivity C-reactive protein (hs-CRP) | 12 weeks
  The change of inflammation indicators before and after intervention.
Vascular endothelial growth factor (VEGF) | 12 weeks
  The change of growth factor indicators before and after intervention.
Insulin-like growth factor(IGF-1) | 12 weeks
  The change of growth factor indicators before and after intervention.
Malondialdehyde (MDA) | 12 weeks
  The change of malondialdehyde (MDA) level before and after intervention.
Superoxide dismutase (SOD) | 12 weeks
  The change of superoxide dismutase (SOD) level before and after intervention.
Nitric oxide (NO) | 12 weeks
  The change of nitric oxide (NO) level before and after intervention.
Heart rate variability (HRV) | 12 weeks
  The change of heart rate variability (HRV) before and after intervention.
Mean flow rate (Vm) of middle cerebral artery and carotid artery | 12 weeks
  The change of middle cerebral artery mean flow rate and carotid artery mean flow rate before and after intervention.
Resistance index (RI) of middle cerebral artery and carotid artery | 12 weeks
  The change of middle cerebral artery resistance index and carotid artery resistance index before and after intervention.
Pulsatility index (PI) of middle cerebral artery and carotid artery | 12 weeks
  The change of middle cerebral artery pulsatility index and carotid artery pulsatility index before and after intervention.
Peak systolic velocity (PSV) and end-diastolic velocity (EDV) of carotid artery | 12 weeks
  The change of peak systolic velocity and end-diastolic velocity of carotid artery before and after intervention.
Vascular endothelial function indicator: Flow-mediated dilation (FMD) | 12 weeks
  The change of flow-mediated dilation before and after intervention.
Artery stiffness indicator: Carotid-femoral pulse artery stiffness (cfPWV). | 12 weeks
  The change of carotid-femoral pulse artery stiffness (cfPWV) before and after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sports Medicine and Rehabilitation, Beijing Sport University, Beijing, China